CLINICAL TRIAL: NCT00510055
Title: The Effect of Subcision and Calcium Hydroxylapatite (Radiesse) Injection on Rolling Acne Scarring Appearance
Brief Title: Treatment of Acne Scarring With a Novel Procedure Combination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology- Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU752
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Acne Scarring
MeSH Terms: interventions — Prolaryn Plus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): scars receive subdermal manipulation ONLY
  Interventions: Procedure: subdermal manipulation ONLY
- B (Experimental): scars receive subdermal manipulation AND injection of a filler
  Interventions: Procedure: subdermal manipulation AND injection of a filler

INTERVENTIONS:
Procedure: subdermal manipulation ONLY — scars receive subdermal manipulation ONLY
  Other Names: subcision
  Arms: A
Procedure: subdermal manipulation AND injection of a filler — scars receive subdermal manipulation AND injection of a filler
  Other Names: Radiesse
  Arms: B

SUMMARY:
The primary objective of this study is to look at the efficacy of subdermal manipulation and filler injection in the improvement of acne scar appearance.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether the use of subcision in conjunction with calcium hydroxylapatite injections will improve the appearance of rolling acne scars better than subcision alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Have two acne scar areas
* The subjects are in good health
* The subject has the willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator.

Exclusion Criteria:

* Under 18 years of age
* Pregnancy or Lactation
* Subjects who are unable to understand the protocol or to give informed consent
* Subjects with mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Scar Improvement | 3.5 months

SECONDARY OUTCOMES:
Adverse Events | 3.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States